CLINICAL TRIAL: NCT06141317
Title: Tissue Regeneration and Function Recovery in Patients With Parkinson's Disease Using Allogenic Pluripotent Stem Cells Isolated From Adipose Tissue (PASCs): A Randomized Phase I/IIa Clinical Trial (REPOSE)
Brief Title: Randomized Clinical Trial in Parkinson's Disease Patients Using Pluripotent Adipose Stem Cells (PASCs)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ClusterXStem-Costa Rica (Other)
Collaborators: Universidad de Costa Rica (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: Pluripotency; Non-tumorigenic; Neurodegenerative disease; Safety; Efficacy; Tissue/function regeneration; Improve symptoms; Potential cure
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PASC transplantation (25 million PASCs/patient) (Experimental): Pluripotent Adipose-Derived Stem Cells will be delivered intravenously
  Interventions: Biological: PASC transplantation (25 million PASCs/patient)
- Control (Placebo Comparator): Saline solution will be delivered intravenously
  Interventions: Biological: Control

INTERVENTIONS:
Biological: PASC transplantation (25 million PASCs/patient) — 3 doses of 25 million PASCs implantation via peripheral vein (Day 0, 3 months, 6 months)
  Arms: PASC transplantation (25 million PASCs/patient)
Biological: Control — 0.9% saline solution via peripheral vein (Day 0, 3 months, 6 months)
  Arms: Control

SUMMARY:
The purpose of this study is to assess the safety and efficacy of allogenic pluripotent stem cells isolated from adipose tissue (PASCs) in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
Pluripotent Adipose-Derived Stem Cells (PASCs) will be delivered intravenously at a dosage of 25 million PASCs/patient to Parkinson's Disease patients for three infusions each spaced 3 months apart (0, 3, and 6 months). Safety and efficacy of PASC treatment will be monitored over 0, 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men ≥18 years of age or women ≥45 years of age
2. Written informed consent
3. Receiving drug treatment for diagnosis of mild to moderate Parkinson's Disease
4. Modified Hoehn and Yahr stage 1, 2, or 3
5. Diagnosed with Parkinson's Disease for more than 5 years
6. Stable treatment regimen that has not been modified in the 90 days prior to the start of the study
7. No expected addition of symptomatic therapy for at least one year after the start of the study
8. Women of reproductive age must use contraceptive treatment

Exclusion Criteria:

1. Drug-induced Parkinsonism
2. Parkinsonism associated with stroke, progressive supranuclear palsy, Lewy body disease, corticobasal degeneration, or multiple system atrophy
3. Major psychiatric comorbidity that prevents ensuring study follow-up
4. History of alcohol or drug use
5. History of brain surgery for Parkinson's Disease
6. Serious complications deemed inappropriate by Principal Investigator
7. Diagnosis of advanced-stage medical conditions (chronic liver injury with Child-Pugh B or higher, chronic obstructive pulmonary disease with Gold C or higher, or heart failure with ejection fraction <35%)
8. Use of cytostatic drugs
9. Patients with life expectancy < 6 months
10. Diabetes mellitus with poor metabolic control (HbA1c > 8%)
11. Active infectious disease requiring medical treatment
12. Use of systemic steroids or immunosuppressive drugs
13. Patients positive for Hepatitis B antigen, Hepatitis C antibody, or HIV antibody
14. Fertile, pregnant, possibly pregnant, or lactating women
15. History of active mesenchymopathies
16. Active malignancy or diagnosis of malignancy in the last 5 years
17. Abnormal laboratory values, including:

    * AST >1.5 times Upper Limit of Normal (ULN) (Normal Range: 8 to 48 Units/L)
    * ALT >1.5 times ULN (Normal Range: 7 to 55 Units/L)
    * Bilirubin >1.5 times ULN (Normal Range: 0.2 to 1.2 mg/dL)
    * Creatinine >1.5 times ULN (Normal Range: 0.5 to 1.30 mg/dL)
    * Hematocrit significantly outside normal range (36% to 54%)
    * Lymphocytes significantly outside normal range (103 to 4.8 x 103 lymphocytes/μL)
    * Monocytes significantly outside normal range (200 to 800 lymphocytes/μL)
    * Neutrophils significantly outside normal range (2.5 x 103 to 7 x 103 lymphocytes/μL)
    * Erythrocytes significantly outside normal range (4.7 x 106 to 6.1 x 106 lymphocytes/μL)
    * Platelets significantly outside normal range (150 x 103 to 450 x 103 lymphocytes/μL)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in motor function as assessed by the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  The MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a widely used research tool to quantify the clinical characteristics of PD in adults. This scale assesses various aspects of Parkinson's disease, including motor and non-motor experiences of daily life and motor complications. This test will take approximately 30 minutes, assessing the impact of the disease in 4 different domains distributed in 65 items, of which 48 are scored from 0 to 4 and seven with dichotomous answers of "yes" or "no". The global range of the MDS-UPDRS will be from 0 to 260 points, the higher the score, the greater the disease involvement.
Quality of life as assessed by the 39-item Parkinson's disease Questionnaire (PDQ-39) | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  The 39-item Parkinson's disease Questionnaire (PDQ-39) is the most widely test used to assess specific quality of life questionnaire for Parkinson's disease, and it has been validated and cross-culturally translated. The questionnaire consists of 39 questions to be completed by the patient, that assesses the frequency in which patients with PD experience difficulties in 8 dimensions of functionality and well-being: mobility, activities of daily living, emotional well- being, attention and memory, social support, depression, cognition, communication and social relationships. Items can be transformed on a linear scale from 0 to 100, the higher the score reflects a lower quality of life.
Speech voice sound and duration | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  Since most people with Parkinson's disease (PD) have voice and speech disorders that result in harmful effects on communication and quality of life; the measurement of the pressure level and sound duration will be executed using the Samson Go Mic and the software used for the Lee Silverman Voice Treatment Therapy (LSVT LOUD).
Dynamic balance and movement during translational motion and single-limb stance in seconds as assessed by the Mini Balance Evaluation Systems Test (mini BESTest) | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  The Mini Balance Evaluation Systems Test (mini BESTest) has proven to be a reliable and valid measurement tool for patients with PD. It is aimed to measure dynamic balance and associated movement during translational motion. The test consists of 14 items, with a maximum score of 28 points, with a higher test result, the greater the patient's functionality 35 . The test has high inter-rater reliability (ICC = 0.92) and high test-retest reliability (ICC = 0.92) for PD patients.
Balance as assessed by the The Five-times Sit-to-stand Test | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  The Five-times sit-to-stand Test is a tool that quantifies the ability of patients suffering from diseases associated with balance problems, as in the case of PD, to perform transitional motions. In addition, it has been used as a measure of lower limb strength. The test has excellent inter-rater reliability and high test-retest reliability, as well as assessing for the risk of falls in patients with PD.
Mobility and fall risk as assessed by the Timed "Up & Go" test | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  The Timed "Up & Go" test consists of observing and timing the patient as he gets up from an armchair, walking for 3 meters, turns, returns and sits down again. The results of this test correlates well with the logarithmic transformation scores on the Berg Balance Scale, gait speed and the Barthel Index of AVD (Activities of Daily Living), and can predict the patient's ability to walk alone safely.
Balance and postural stability as assessed by the Clinical test of Sensory Interaction & Balance Test (CTSIB), stability limits, and unipodal balance test | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  Computerized posturography using a force platform system provides objective and quantitative evaluations of deficiencies in postural control. The participants of the present study will be subjected to two tests of balance and postural stability using the HUMAC®43 brand force platform system. Three tests will be performed: CTSIB test (Clinical test of Sensory Interaction & Balance), the stability limits, and the unipodal balance test.
Tremor and handwriting | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  Alterations in the kinematics of handwriting are among the recently proposed biomarkers of PD. Recent studies have suggested the potential of handwriting analysis for both early diagnosis and assessment of disease progression. In the present study, the patients will be subjected to 5 tests, at 5 different times of the study using the MovAlyzeR® software in conjunction with the WACOM ONE tablet, to measure the speed, amplitude, fluidity and tremor of the movements of the upper extremities.
Grip strength | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  The decrease in grip strength is a predictor of adverse outcomes in older adults and will be determined using a Jamar brand digital dynamometer to measure the grip strength of the patients participating in each assessment.
Dynamic balance in the bipedal as measured by the 360 degree turn test | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  This test measures dynamic balance in the bipedal. In this test, the number of steps and the time that take the patient to make a complete 360-degree turn will be measured.

SECONDARY OUTCOMES:
Adverse events upon clinical examination | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  Study participants will be examined for clinical signs of adverse events.
Optimal number of doses of 2.5 x 10^7 PASCs for therapeutic response | Day 0, 1 Month, 3 Months, 6 Months, 12 Months
  The optimal number of doses of PASCs for therapeutic response will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Henriquez, M.D., Principal Investigator — Hospital Clínica Católica
Locations (2):
- Costa Rica (2):
  - Hospital Clínica Católica, San José
  - Clínica NeuroFT, San José

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heneidi S, Simerman AA, Keller E, Singh P, Li X, Dumesic DA, Chazenbalk G. Awakened by cellular stress: isolation and characterization of a novel population of pluripotent stem cells derived from human adipose tissue. PLoS One. 2013 Jun 5;8(6):e64752. doi: 10.1371/journal.pone.0064752. Print 2013. PMID 23755141
- [Background] Gimeno ML, Fuertes F, Barcala Tabarrozzi AE, Attorressi AI, Cucchiani R, Corrales L, Oliveira TC, Sogayar MC, Labriola L, Dewey RA, Perone MJ. Pluripotent Nontumorigenic Adipose Tissue-Derived Muse Cells have Immunomodulatory Capacity Mediated by Transforming Growth Factor-beta1. Stem Cells Transl Med. 2017 Jan;6(1):161-173. doi: 10.5966/sctm.2016-0014. Epub 2016 Aug 2. PMID 28170177
- [Background] Simerman AA, Phan JD, Dumesic DA, Chazenbalk GD. Muse Cells: Nontumorigenic Pluripotent Stem Cells Present in Adult Tissues-A Paradigm Shift in Tissue Regeneration and Evolution. Stem Cells Int. 2016;2016:1463258. doi: 10.1155/2016/1463258. Epub 2016 Dec 14. PMID 28070194
- [Background] Fisch SC, Gimeno ML, Phan JD, Simerman AA, Dumesic DA, Perone MJ, Chazenbalk GD. Pluripotent nontumorigenic multilineage differentiating stress enduring cells (Muse cells): a seven-year retrospective. Stem Cell Res Ther. 2017 Oct 18;8(1):227. doi: 10.1186/s13287-017-0674-3. PMID 29041955
- [Background] Yamashita T, Kushida Y, Abe K, Dezawa M. Non-Tumorigenic Pluripotent Reparative Muse Cells Provide a New Therapeutic Approach for Neurologic Diseases. Cells. 2021 Apr 20;10(4):961. doi: 10.3390/cells10040961. PMID 33924240
- [Background] Leung KL, Chazenbalk GD. Human Pluripotent Nontumorigenic Multilineage Differentiating Stress Enduring (Muse) Cells Isolated from Adipose Tissue: A New Paradigm in Regenerative Medicine and Cell Therapy. In Scientific Principles of Adipose Stem Cells, edited by: L Kokai, K Marra, JP Rubin, Editorial Elsevier, Chapter 6, 91-108, 1st Edition, 2021, https://doi.org/10.1016/B978-0-12-819376-1.00004-4
- See also: Patent: Pluripotent human adipose adult stem cells: isolation, characterization and clinical implications — http://patents.google.com/patent/WO2014190150A1/un